CLINICAL TRIAL: NCT02843750
Title: A Pilot Study of Inspiratory Muscle Training for Patients Undergoing Esophageal Surgery
Brief Title: Study of Inspiratory Muscle Training for Patients Undergoing Esophageal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-009190
Record Dates: First submitted 2016-07-11; First posted 2016-07-26 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Cancer of Esophagus; Cancer of the Esophagus; Esophageal Cancer; Esophagus Cancer; Esophagus Neoplasm; Neoplasms, Esophageal
Keywords: Rehabilitation; Inspiratory Muscle Training
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inspiratory Muscle Training-Rehabilitation (Experimental): Patients will start the IMT-R, following their consent and within 2 weeks of their scheduled surgery: 10 sessions lasting about 90 minutes. Participants who completed their initial IMT greater than 2 weeks prior to surgery will have an additional visit prior to surgery. Participants will receive a Participant Manual demonstrating and explaining the rehabilitation process. Participants will also receive a log for recording their efforts and notes. A DVD of the rehabilitation is available to the participant. Participants will complete questionnaires at baseline and 3 months.
  Interventions: Behavioral: Inspiratory Muscle Training-Rehabilitation; Other: Questionnaires

INTERVENTIONS:
Behavioral: Inspiratory Muscle Training-Rehabilitation — The training will include the following components:
  1. Breathing Awareness
  2. Upper and Lower Extremity Exercise.
  3. Instructions for Inspiratory Muscle Training (IMT) performed using the PFlex valve
  4. Practice at home
Other: Questionnaires — Patient quality of life will be measured using patient-reported outcomes measurement information system (PROMIS) global items. Patients will also complete the Chronic Respiratory Questionnaire (CRQ) and the Medical Research Council Dyspnea Scale (MCR).

SUMMARY:
To obtain definitive evidence for the effectiveness of a short preoperative inspiratory muscle training (IMT) protocol on the morbidity and recovery from an esophageal surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with esophageal cancer and scheduled for esophageal resection at the Mayo Clinic Rochester with gastric conduit reconstruction -Cognitively capable to understand and perform a preoperative program
* Able to follow the intervention program for at least 2 weeks before surgery (surgery is usually scheduled 4 to 12 weeks after radiation)
* Willing to sign the informed consent form

Exclusion Criteria:

* Unable to communicate in the English language
* Participating in a conflicting trial concerning esophageal resection

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pneumonia | 3 months
  To prospectively determine the effect of a customized preoperative inspiratory muscle training (IMT) and brief pulmonary rehabilitation program on the incidence of postoperative pneumonia in patients that undergo an esophageal surgical resection. The investigators will consider the following as pneumonia: new infiltrate + either fever (>38.5 C) and white cell count >11,000 or fever and purulent secretions.

SECONDARY OUTCOMES:
Postoperative Pulmonary Complications | 3 months
  To prospectively determine the effect of a customized preoperative inspiratory muscle training (IMT) and brief pulmonary rehabilitation program on the incidence of postoperative pulmonary complications in patients that undergo an esophageal surgical resection.The investigators will consider the following events as post-operative pulmonary complications: severe atelectasis (requiring bronchoscopy) and respiratory failure (intubation or prolonged mechanical ventilation (>24hours).

OTHER OUTCOMES:
Length of Hospital Stay | 3 months
  Length of hospital stay will be measured by participant monitoring while hospitalized until hospital discharge.
Quality of Life | Baseline to 3 months
  Quality of life will be assessed at baseline and at 3 months after hospital discharge by participant completion of the PROMIS Global 10.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No